CLINICAL TRIAL: NCT07041320
Title: Effect and Safety of Oral Metronomic Vinorelbine and PD-1 Inhibitors in Elderly Patients With Non-small Cell Lung Cancer
Brief Title: Oral Metronomic Vinorelbine and PD-1 Inhibitors in Elderly Non-small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Anhui Chest Hospital (Other)
Responsible Party: Principal Investigator, Guan Maojing, Associate chief physician, Anhui Chest Hospital
Other Study IDs: Anhui Chest Hospital
Record Dates: First submitted 2025-03-31; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer (NSCLC); Elderly (People Aged 65 or More)
Keywords: Oral metronomic vinorelbine; PD-1 inhibitors
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The goal of this observational study is to evaluate the efficacy and safety of oral metronomic vinor: Participants over 65 years old, received oral metronomic vinorelbine 40mg every week (20mg for patients over 80 years old), combined with PD-1 inhibitors every 3 weeks.

SUMMARY:
The goal of this observational study is to evaluate the efficacy and safety of oral metronomic vinorelbine and PD-1 inhibitors in elderly patients with unoperable, locally advanced or metastatic non-small-cell lung cancer. The primary end point was objective response rate (ORR), and the second end points included disease control rate (DCR), progression-free survival (PFS), and safety. Participants over 65 years old, received oral metronomic vinorelbine 40mg every week (20mg for patients over 80 years old), combined with PD-1 inhibitors every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1) All patients are histologically or cytologically confirmed non-small cell lung cancer. Genetic testing identifies no driver gene mutations.

  2) Male or female, age ≥ 65 years 3) Patients had not received first-line treatment. 4) KPS score ≥ 70 points (ECOG score 0-1 points), the expected survival ≥3 months; 5) No dysfunction of major organs. EcG, liver function, renal function, and blood count tests before treatment are normal or basically normal, but must meet the following experimental results:
  1. Blood routine test:

     Leukocyte WBC≥3.5×109/L; Neutrophil count (ANC) ≥ 1.5×109/L; Platelet (PLT) ≥ 80×109/L;
  2. Blood biochemical test:

     Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal values; Alanine aminotransferase (ALT/SGPT) and alanine transaminases (AST/SGOT) ≤ 2.5 times the normal high value (ULN), or ≤ 5 times the upper limit of normal value in patients with liver metastases; Serum creatinine (Cr) ≤ 1.5 times the upper limit of normal values;
  3. Cardiac function test: 50% of the left ventricular ejection function of the heart >; 6) The subject has good compliance, and can cooperates with follow-up.

     Exclusion Criteria:
* previously treated

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years old with unoperable, locally advanced or metastatic non-small-cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) | at the end of every 2 cycles(each cycle is 21 days),through study completion, an average of 2 years
  CR+PR/All patients(%)

SECONDARY OUTCOMES:
disease control rate (DCR) | at the end of every 2 cycles(each cycle is 21 days),through study completion, an average of 2 years
  CR+PR+SD/All patients(%)
progression-free survival (PFS) | at the end of every 2 cycles(each cycle is 21 days),through study completion, an average of 2 years
  PFS was calculated from treatment initiation to disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Qingming Shi, Doctor, Principal Investigator — Anhui Chest Hosptial
Locations (1):
- Anhui Chest Hosptial, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No